CLINICAL TRIAL: NCT06741046
Title: Evaluation of the Treatment Response and Prognosis of Cervical Adenocarcinoma/adenosquamous Carcinoma After Radiotherapy: a Retrospective Study
Brief Title: RT for Cervical Adenocarcinoma/adenosquamous Carcinoma
Status: Active, not recruiting | Type: Observational
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Principal Investigator, yanjunfang, Chief Assistant for Department of Radiotherapy, Peking Union Medical College Hospital
Other Study IDs: ATTRACT-Retro
Record Dates: First submitted 2024-12-16; First posted 2024-12-18 (Actual); Last update posted 2024-12-18 (Actual); Status verified 2024-11

CONDITIONS: Uterine Neoplasms; Genital Neoplasms, Female
Keywords: cervical adenocarcinoma; cervical adenosquamous carcinoma
MeSH Terms: conditions — Uterine Neoplasms; Genital Neoplasms, Female

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — biopsy
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Radical surgery group: Patients who received radical surgery for cervical cancer in Peking Union Medical College Hospital
- Concurrent chemoradiotherapy group: Patients who received concurrent chemoradiotherapy in Peking Union Medical College Hospital

SUMMARY:
The purpose of this study was to retrospectively analyze patients with cervical adenocarcinoma/adenosquamous carcinoma who had been admitted to our hospital. Approximately 500 cases of cervical adenocarcinoma were planned to be included, summarize the disease characteristics, treatment regimens, and recurrence patterns of the patients, and analyze the association between treatment regimens and recurrence patterns and prognosis.

DETAILED DESCRIPTION:
This study is a retrospective analysis. The keywords "cervical adenocarcinoma" and "cervical adenosquamous carcinoma" were used to search for patients with cervical adenocarcinoma and cervical adenosquamous carcinoma admitted to the Department of Radiotherapy, Peking Union Medical College Hospital from 2009 to 2024. The clinical information, pathological information, and treatment methods of the patients in the medical records were collected, and the date of death, cancer recurrence, and metastasis were confirmed by querying medical records or conducting telephone interviews. The included cases were divided into the radical surgery group and the concurrent chemoradiotherapy group according to the treatment mode. The pathological types were reclassified according to the IECC 2018 standards, and the associations between pathological types, treatment regimens, recurrence patterns (local recurrence, distant metastasis, recurrence within the irradiation field, recurrence outside the irradiation field), and prognosis were analyzed. For patients with residual local cervical tumors after synchronous chemoradiotherapy or recurrence within the field after radiotherapy, the previous genetic test results of the patients were retrieved, their genomic characteristics were analyzed, and compared with the TCGA database. If the patient has not undergone genetic testing before, pathological sections of the patient will be obtained from our hospital for whole exome sequencing, and the testing items include.

ELIGIBILITY:
Inclusion Criteria:

a) Pathological diagnosis of cervical adenocarcinoma; b) Age 18-80 years old; c) Karnofsky score≥60 points; e) Complete blood count, and comprehensive metabolic panel meet the conditions for CCRT or RT after surgery; f) No metal implants in the body, and can perform MRI examination; g) Willing to participate in this study and provide written informed consent. -

Exclusion Criteria:

1. Patients who have received pelvic radiotherapy before;
2. Patients whose target tumors have been treated before (chemotherapy, immunotherapy, surgical treatment, etc.);
3. Allergy to iodine contrast agent;
4. Participating in other clinical studies that may affect the results of this study (determined by the principal investigator);

f) Serious diseases that may significantly affect compliance with clinical trials, such as unstable heart disease, kidney disease, chronic hepatitis, poorly controlled diabetes, and mental illness that require treatment; g) Other situations that the investigator believes are not suitable for participation in this clinical study.

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Female patinets diagnosed with cervical adenocarcinoma or adenosquamous carcinoma receiving CCRT or RT after complete surgery
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2014-06-01 (Actual); Primary Completion 2025-06-01 (Estimated); Study Completion 2027-06-01 (Estimated)

PRIMARY OUTCOMES:
Local control rate | local control rates at 2 years or 3 years after the initial treatment
  Tumor control rate in the cohort after treatment

SECONDARY OUTCOMES:
Progress free survival | 2 years after initial treatment
  the time from initial treatment to disease progression or death from any cause.
Overall survival | 2 years after initial treatment
  The length of time from the start of initial treatment to death or the last followup

CONTACTS AND LOCATIONS:
Locations (1):
- Peking Union Medical College Hospital, Beijing, China